CLINICAL TRIAL: NCT06276491
Title: A Phase 1, First-in-Human, Dose Escalation and Expansion Study to Evaluate the Safety and Tolerability of XmAb541 in Advanced Solid Tumors
Brief Title: Phase 1, Safety and Tolerability Study of XmAb541 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XmAb541-01
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Germ Cell Tumor; Testicular Germ Cell Tumor; Ovarian Germ Cell Tumor
Keywords: Phase 1; Ovarian Cancer; CLDN6; Testicular Cancer; Germ Cell Tumor; Endometrial Cancer; T-cell Engager
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Neoplasms, Germ Cell and Embryonal; Testicular Germ Cell Tumor; Testicular Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation and Dose Expansion of XmAb541 (Experimental): Intravenous or Subcutaneous administration
  Interventions: Biological: XmAb541

INTERVENTIONS:
Biological: XmAb541 — Monoclonal bispecific antibody

SUMMARY:
The primary purpose of this study is to determine whether the investigational drug XmAb541 is safe and well tolerated, and to determine an optimal and safe dose(s) for further study. The study will also evaluate the effect of XmAb541 on tumor outcomes.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years. For subjects with GCTs, age ≥15 years
* CLDN6+ tumor
* Histological or cytological documentation of locally advanced, recurrent, or metastatic ovarian, fallopian tube, or peritoneal cancer, adenocarcinoma of the endometrium (endometrial cancer, uterine cancer, or carcinoma of the uterine corpus), GCT
* Have documented progressive disease (PD) on standard-of-care therapies appropriate for the specific tumor type; have exhausted therapies with a survival benefit or the standard therapy has no survival benefit or proven to be ineffective, intolerable, or subject is not a candidate for such available therapy.
* Eastern Cooperative Oncology Group performance status of 0-2
* Life expectancy ≥ 3 months
* Adequate liver, kidney, and bone marrow function

Key Exclusion Criteria:

* Prior exposure to a CLDN6 targeting product
* Ovarian cancer that is platinum refractory, or has rapid progression on most recent prior ≥ second line systemic anticancer therapy
* Have known active central nervous system metastases and/or carcinomatous meningitis. Patients with treated brain metastases may participate, provided they are radiologically stable.
* Active known or suspected autoimmune disease
* Have any condition requiring systemic treatment with corticosteroids, prednisone equivalents, or other immunosuppressive medications within 14 days prior to first dose of study drug
* Clinically significant cardiovascular, pulmonary or gastrointestinal disease
* Positive test for hepatitis C RNA
* Positive test for hepatitis B surface antigen or hepatitis B core antibody (hBcAb)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Day 1 to 2 years
Incidence of dose-limiting toxicities (DLTs) | Day 1 to Day 28
Incidence of cytokine release syndrome (CRS) | Day 1 to Day 28

SECONDARY OUTCOMES:
Measurement of Cmax | Day 1 to 2 years
  Peak plasma concentration
Measurement of area under curve (AUC) | Day 1 to 1.4 years
  Area under the plasma concentration versus time curve
Measurement of Ctrough | Day 1 to 2 years
  Plasma concentration before next dose
Objective Response Rate | Day 1 to 2 years
  Objective Response Rate by RECIST 1.1 assessment of CT/MRI imaging
Duration of Response | Day 1 to 2 years
  Duration of Response Objective Response Rate by RECIST 1.1 assessment of CT/MRI imaging
Changes in Circulating Tumor DNA (ctDNA) | Day 1 to 2 years
  Maximum variant frequency or mean/median variant frequency

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Karmanos Cancer Institute, Detroit, Michigan
  - The John Theruer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Einstein Comprehensive Cancer Center, The Bronx, New York
  - The Ohio State University, Columbus, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - SCRI Oncology Partners, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia